CLINICAL TRIAL: NCT05585996
Title: Exploratory Clinical Study of CD19-targeted CAR-T and CAR-DC in the Treatment of Relapsed and Refractory B-cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0160
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Relapsed and Refractory B-cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination therapy of CD19 CAR-T and CD19 CAR-DC (Experimental): 6-18 patientsare planned to be enrolled in the dose-escalation trial (0.5×10^6/kg、1×10^6/kg、2×10^6/kg和4×10^6/kg) and 52 patients in the dose-expansion trial.
  Interventions: Biological: CD19 CAR-T and CD19 CAR-DC

INTERVENTIONS:
Biological: CD19 CAR-T and CD19 CAR-DC — Intravenously injected CAR DC cells and followed by CAR T cells 4 hours later

SUMMARY:
This is an open, single-arm, prospective, dose-escalation clinical trial designed to evaluate the safety and the preliminary efficacy of CD19-targeted CAR-T combined with CAR-DC in the treatment of relapsed and refractory B-cell lymphoma

DETAILED DESCRIPTION:
6-18 patients are planned to be enrolled in the dose-escalation trial. The dose of CD19-CAR-DC was according to the 3+3 dose-escalation principle (0.25×10^6/kg, 0.5×10^6/kg, 0.75×10^6/kg ( ±20%) . CAR-T was 2×10^6/kg . The primary endpoints are DLT, MTD, and the second endpionts are the overall response rates (CR and PR), overall survival, and progression-free survival. Based on the results in the dose-escalation trial, the recommended dose will be determined. Another 52 patients will be enrolled to continue estimating the safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18 to 75 years old at the time enrollment, with ECOG Score of ≤ 3;
2. Patients should provide a written informed consent;
3. Histologically confirmed CD19+ DLBCL, HGBL-DHL, MCL, tFL, PMBL;

   * Confirmation obtained from central pathology review before enrollment;
   * Sufficient formalin-fixed, paraffin-embedded tumor samples were required for histologically confirmed diagnosis and detection of CD19 expression;
   * Relapsed DLBCL and tFL after ≥2 lines of chemotherapy that include rituximab and anthracycline, or refractory disease as defined in the SCHOLAR-1 study: progressive disease after receiving ≥ 4 cycles of first-line therapy or stable disease (received 2 cycles of later-line therapy) as best response to chemotherapy or relapse ≤ 12 months after autologous stem cell transplantation (ASCT);
   * Relapsed/refractory MCL after ≥ 2 lines of prior therapy, including immunochemotheapy and BTK inhibitor such as ibrutinib, or patient did not agree to receive BTK inhibitor treatment;
   * At least one measurable tumor according to revised International Working Group (IWG) Response criteria;
4. Life expectancy ≥ 3 months;
5. Adequate cardiac, pulmonary, liver, renal, and bone marrow functions, with the following laboratory values: an absolute neutrophil count > 1,000/mm3, platelets count ≥ 45,000/mm3, and hemoglobin > 8.0g/dl; alanine aminotransferase and aspartate aminotransferase ≤ 2.5 × the upper limit of the normal range (ULN), and total bilirubin ≤ 2.0 mg/dl; a serum creatinine of ≤ 1.5 × ULN; a left ventricular ejection fraction ≥ 50%;

Exclusion Criteria:

1. Prior treatment that included anti-CD19-targeted therapy, CAR T cell therapy, gene therapy, and allogenic hematopoietic stem cell transplantation (allo-HSCT);
2. Chemotherapy other than lymphodepleting chemotherapy, therapeutic doses of steroids, immunosuppressive agent, any radiation therapy or anti-tumor targeted therapy including lenalidomide, bortezomib, ibrutinib, received within 2 weeks before cell collection;
3. Clinical trial with investigational drug was performed within 4 weeks;
4. History of other cancers;
5. Active hepatitis B or hepatitis C. Hepatitis B: HBV-DNA ≥ 1,000 IU/ml; Hepatitis C: HCV RNA positive;
6. HIV infection;
7. Uncontrollable infection of active bacteria and fungi;
8. Currently pregnant or refusal to practice birth control within 1 year;
9. Active autoimmune or inflammatory diseases;
10. Central nervous system lymphoma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-75 years
Enrollment: 70 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
DLT | Up to 28 days
  To evaluate the safety, tolerability, and determine the recommended dosage of combined therapy of CD19 CAR-T and CD19 CAR-DC for Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
MTD | Up to 28 days
  MTD was the highest dose for DLT in ≤1/6 subjects
Incidence of abnormalities | Up to 28 days
  Incidence of abnormalities in AE/SAE/AESI/laboratory tests/electrocardiograms/vital signs.

SECONDARY OUTCOMES:
Overall Response Rate | Up to 2 years
  The proportion of CR or PR patients as assessed by investigators based on Lugano 2014 Response Assessment
Duration of Response | Up to 2 years
  The time from the start of the first assessment of CR or PR to the first assessment as disease recurrence or progression or death
Progression Free Survival | Up to 2 years
  The length of time that a participant's disease did not progress during or after CAR-T treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Qian, MD, PhD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang Universit
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No